CLINICAL TRIAL: NCT00154141
Title: A Prospective, Randomized Controlled Study to Compare the Effects of a Fibrin Sealant (FS2) Versus Manual Compression on Haemostatic Efficacy During Vascular Surgical Procedures Utilising Polytetrafluorethylene Graft Material on an End-to-Side Femoral or Upper Extremity Vascular Access Arterial Anastomosis
Brief Title: Evaluation of Fibrin Sealant 2 in Vascular Surgical Procedures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Collaborators: OMRIX Biopharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 400-05-001
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2006-07-13 (Estimated); Status verified 2006-07

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Fibrin Tissue Adhesive

INTERVENTIONS:
Drug: Fibrin sealant (FS2)

SUMMARY:
A comparison of a fibrin sealant versus manual compression in stopping surgical bleeding during vascular procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, 18 years or older, requiring elective, primary or repeat vascular procedures with at least one end-to-side femoral or upper extremity vascular access arterial anastomosis (e.g. femoral-femoral, femoral-popliteal, femoral-tibial, ilio-femoral, aorto-bifemoral, abdominal aortic aneurysm, upper extremity vascular access for dialysis) using uncoated or heparin-coated PTFE grafts and polypropylene sutures (size 5-0 or 6-0) with a 1:1 needle-to-thread ratio.
* Following initial arterial clamp release, the study surgeon determines that adjunctive measures are needed to obtain haemostasis at the SAS.
* Subjects must be willing to and capable of participating in the study, and provided written informed consent.

Exclusion Criteria:

* Subjects undergoing re-vascularisation using autologous conduits (e.g. saphenous vein) or prosthetic material other than uncoated or heparin-coated PTFE.
* Subjects undergoing emergency surgery.
* Subjects with any intra-operative findings that may preclude conduct of the study procedure.
* Subjects with known intolerance to heparin, blood products or to one of the components of the study product.
* Subjects unwilling to receive blood products.
* Subjects with autoimmune immunodeficiency diseases (including known HIV).
* Subjects who are known, current alcohol and / or drug abusers.
* Subjects who have participated in another investigational drug or device research study within 30 days of enrolment.
* Female subjects who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2005-06; Study Completion 2006-03

PRIMARY OUTCOMES:
Attainment of hemostasis at following randomization.

SECONDARY OUTCOMES:
Attainment of hemostasis following randomization.
Incidence of treatment failures
Incidence of potential bleeding-related complications
Adverse events

CONTACTS AND LOCATIONS:
Locations (17):
- United States (13):
  - Baptist Medical Center, Jacksonville, Florida
  - Memorial Hospital, Jacksonville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Iowa Heart Center, Des Moines, Iowa
  - Univ of Mass Medical Center, Worcester, Massachusetts
  - Hackensack Medical Center, Hackensack, New Jersey
  - Alband Medical Center, Albany, New York
  - Millarad Fillmore Hospital, SUNY, Buffalo, New York
  - Jobst Vascular Center, Toledo, Ohio
  - Vanderbilt Univ Medical Center, Nashville, Tennessee
  - UVA Health System, Charlottesville, Virginia
  - Vascular and Transplant Specialists, Norfolk, Virginia
- United Kingdom (4):
  - Aberdeen Royal Infirmary, Aberdeen
  - Birmingham Heartlands Hospital, Birmingham
  - Royal Infirmary of Edinburgh, Edinburgh
  - Hull Royal Infirmary, Hull

REFERENCES:
- [Derived] Ma GW, Kucey A, Tyagi SC, Papia G, Kucey DS, Varcoe RL, Forbes T, Neville R, Dueck AD, Kayssi A. The role of sealants for achieving anastomotic hemostasis in vascular surgery. Cochrane Database Syst Rev. 2024 May 2;5(5):CD013421. doi: 10.1002/14651858.CD013421.pub2. PMID 38695613
- [Derived] Chalmers RT, Darling Iii RC, Wingard JT, Chetter I, Cutler B, Kern JA, Hart JC. Randomized clinical trial of tranexamic acid-free fibrin sealant during vascular surgical procedures. Br J Surg. 2010 Dec;97(12):1784-9. doi: 10.1002/bjs.7235. Epub 2010 Aug 20. PMID 20730858